CLINICAL TRIAL: NCT04005573
Title: Assessing the Combined Effect of Omega-3 Fatty Acid and Vitamin D3 on Lipid Profile Levels and Oxidized Low Density Lipoprotein: a Randomized Controlled Trial in Males and Females With Vitamin D Deficiency
Brief Title: The Combined Effect of Omega-3 Fatty Acid and Vitamin D3 on Lipid Profile Levels and Oxidized Low Density Lipoprotein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science Private University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DRGS-2014-2015-165-2
Record Dates: First submitted 2019-07-01; First posted 2019-07-02 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-07

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D3; Vitamin D Deficiency; Lipid profile; oxidized low density Lipoprotein; omega-3 fatty acids
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VD3 group (Experimental): dietary supplement : VD3 group treated with 50000 IU VD3/ week for 8 weeks
  Interventions: Dietary Supplement: VD3
- omega 3- FA group (Experimental): dietary supplement : omega 3- FA group 1000 mg wild salmon and fish oil complex (contain 300 mg of omega 3-FA) once daily for 8 weeks
  Interventions: Dietary Supplement: omega 3- FA
- VD3 and omega 3 FA group (Experimental): dietary supplement : VD3 and omega-3FA 50000 IU VD3/week for 8 weeks and 1000 mg wild salmon and fish oil complex (contain 300 mg of omega 3-FA) once daily for 8 weeks
  Interventions: Dietary Supplement: VD3 and omega- 3FA
- control group (Other): no intervention was given
  Interventions: Other: no intervention

INTERVENTIONS:
Dietary Supplement: VD3 — VD3 50000 IU/ week for 8 weeks
  Arms: VD3 group
Dietary Supplement: omega 3- FA — Omega 3 FA group 300 mg once daily for 8 weeks
  Arms: omega 3- FA group
Dietary Supplement: VD3 and omega- 3FA — 50000 IU VD3/week for 8 weeks and 300 mg of omega- 3 FA once daily for 8 weeks
  Arms: VD3 and omega 3 FA group
Other: no intervention — no intervention is given
  Arms: control group

SUMMARY:
The combined effect of omega-3 fatty acid and vitamin D3 on lipid profile levels and oxidized low density lipoprotein: a randomized controlled trial in males and females with vitamin D deficiency

DETAILED DESCRIPTION:
Nothing is published in the literature about the combined effect of vitamin D3 (VD3) and omega-3 fatty acids (omega-3FA) on on lipid profile levels and oxidized low density lipoprotein

This study will be conducted to investigate effect of VD3 and omega-3FA alone and with each other on lipid profile levels and oxidized low density lipoprotein in Jordanian people with vitamin D deficiency.

This randomized, controlled clinical trial will be designed to test effects of 50,000 IU VD3 weekly and 300 mg omega-3FA daily for eight weeks, separately and with each other, on on lipid profile levels and oxidized low density lipoprotein

ELIGIBILITY:
Inclusion Criteria:

* Jordanian people aged 25-55 medical diagnosis of vitamin D deficiency ( VD <25 ng/ ml)

Exclusion Criteria:

* Subjects with previously diagnosed with any chronic disease (cardiovascular disease, osteoporosis, cancer, kidney disease, endocrine disorder, thalassemia) or has a documented history of allergic reactions to n-3FA supplementations

Ages: 22 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
VD 3 | 8 weeks
  Serum level of 25-hydroxyvitamin D
Total Cholesterol | 8 weeks
  serum level of total cholesterol
HDL Cholesterol | 8 weeks
  serum level of HDL Cholesterol
LDL Cholesterol | 8 weeks
  serum level of LDL Cholesterol
triglycerides | 8 weeks
  serum level of triglycerides
oxidized LDL | 8 weeks
  serum level of oxidized LDL

SECONDARY OUTCOMES:
PTH | 8 weeks
  serum level of PTH
Calcium and Phosphorus | 8 weeks
  serum level of Calcium and Phosphorus

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S Abu-Samak, PhD, Principal Investigator — Applied science university
Locations (1):
- Applied Science University, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underline results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: when summary data will published
Access Criteria: open access

REFERENCES:
- [Background] Manson JE, Bassuk SS, Lee IM, Cook NR, Albert MA, Gordon D, Zaharris E, Macfadyen JG, Danielson E, Lin J, Zhang SM, Buring JE. The VITamin D and OmegA-3 TriaL (VITAL): rationale and design of a large randomized controlled trial of vitamin D and marine omega-3 fatty acid supplements for the primary prevention of cancer and cardiovascular disease. Contemp Clin Trials. 2012 Jan;33(1):159-71. doi: 10.1016/j.cct.2011.09.009. Epub 2011 Oct 2. PMID 21986389